CLINICAL TRIAL: NCT02076464
Title: Using Technology to Improve Eating Disorders Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Stanford University (Other)
Responsible Party: Principal Investigator, Denise Wilfley, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01MH100455 (NIH); 5R01MH100455 (NIH)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- StudentBodies - Eating Disorders (Experimental): Participants will participate in the StudentBodies - Eating Disorders program
  Interventions: Behavioral: StudentBodies - Eating Disorders
- Usual Care (No Intervention): Participants will be referred to treatment per protocol at students' corresponding college's mental health services center

INTERVENTIONS:
Behavioral: StudentBodies - Eating Disorders — The intervention is a structured, cognitive-behavioral guided self-help program, derived from manual-based cognitive-behavioral therapy. The intervention targets the core eating disorder pathology (e.g., extreme dietary restraint, overvaluation of shape and weight, binge eating, compensatory behaviors), focusing on helping users develop regular eating patterns, self-control strategies, problem-solving skills, and relapse prevention tools for maintenance of behavior change. The program includes daily symptom checklists, journal exercises and activities, and an asynchronous moderated online discussion group.
  Arms: StudentBodies - Eating Disorders

SUMMARY:
The purpose is to evaluate a technologically-enhanced, guided self-help program to reduce eating disorder outcomes in college-age women.

DETAILED DESCRIPTION:
Colleges are faced with an elevated prevalence of eating disorders, yet less than 20% of students report receiving treatment. Inadequacies in mental health care delivery result in prolonged illness, disease progression, poorer prognosis, and greater likelihood of relapse, highlighting the need for improved modalities for screening and intervention. Over the past 20 years, we have developed a comprehensive, online platform through which we identify and offer tailored evidence-based interventions to individuals across the eating disorder risk and diagnostic spectrum, using minimal person-based resources. The newest intervention in our suite of programs, Student Bodies-Eating Disorders (SB-ED), has not yet been tested in a large-scale trial or via platform delivery. The aim of this study is to conduct the first national deployment of our comprehensive platform and demonstrate that our transdiagnostic guided self-help program, SB-ED, yields measurable and significant improvements in access, costs, and outcomes for eating disorder treatment over referral to usual care (i.e., treatment per protocol at students' corresponding college's mental health services center).

Twenty-eight colleges will be randomly assigned to receive either SB-ED or referral to usual care. We will enroll at least 650 students from these campuses who screen positive for a DSM-5 clinical or subclinical eating disorder (excluding anorexia nervosa, which warrants more intensive medical monitoring). Outcomes will be measured at 6-months, 1-year, and 2-years following the completion of the online screen.

ELIGIBILITY:
Inclusion Criteria:

* Student at a participating college or university ages 18-30
* Screen positive for DSM-5 bulimia nervosa, binge eating disorder, or a subclinical eating disorder

Exclusion Criteria:

* Screen positive for DSM-5 anorexia nervosa
* No access to the internet
* Acutely suicidal

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 690 (Actual)
Dates: Start 2014-01-12 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Change in eating disorder symptoms | Measured at baseline, 6-months, 1-year, and 2-years
  Eating disorder outcomes will be measured using the Eating Disorder Examination Questionnaire

SECONDARY OUTCOMES:
Realized treatment access | 2 years
  Realized treatment access is defined as receipt of eating disorder treatment and will be measured using medical records (when available) and a Health Care Utilization Questionnaire
Eating disorder behavior abstinence rates | 2 years
  Rates of bingeing and purging will be measured using the Eating Disorder Examination Questionnaire
Comorbid symptom severity and impairment | 2 years
  Symptom Severity includes depression, anxiety, alcohol use, eating disorder associated clinical impairment, and academic impairment. These symptoms will be measured using the Patient Health Questionnaire, the PROMIS anxiety questionnaire, an assessment of binge drinking, the Counseling Center Assessment of Psychological Symptoms, the Clinical Impairment Assessment, and academic transcripts (when available).
Service and implementation costs | up to 5 years
  Service and implementation costs will be assessed based on published rates.

CONTACTS AND LOCATIONS:
Overall Officials: Denise E. Wilfley, Ph.D., Principal Investigator — Washington University School of Medicine; C. Barr Taylor, M.D., Principal Investigator — Stanford University

REFERENCES:
- [Derived] Graham AK, Fitzsimmons-Craft EE, Sadeh-Sharvit S, Balantekin KN, Eichen DM, Firebaugh ML, Goel NJ, Monterubio GE, Karam AM, Flatt RE, Jo B, Jacobi C, Wilfley DE, Taylor CB, Trockel M. Moderators and mediators of a digital cognitive behavior therapy-guided self-help intervention for eating disorders: Informing future design efforts. J Consult Clin Psychol. 2023 May;91(5):280-284. doi: 10.1037/ccp0000786. Epub 2023 Jan 12. PMID 36634022
- [Derived] Fitzsimmons-Craft EE, Taylor CB, Graham AK, Sadeh-Sharvit S, Balantekin KN, Eichen DM, Monterubio GE, Goel NJ, Flatt RE, Karam AM, Firebaugh ML, Jacobi C, Jo B, Trockel MT, Wilfley DE. Effectiveness of a Digital Cognitive Behavior Therapy-Guided Self-Help Intervention for Eating Disorders in College Women: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2015633. doi: 10.1001/jamanetworkopen.2020.15633. PMID 32865576